CLINICAL TRIAL: NCT05094427
Title: Perioperative Local Anesthesia Block in Spine Surgery: A Retrospective Chart Review
Brief Title: Perioperative Local Anesthesia Block in Spine Surgery
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAT6085
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Spine Disease; Lumbar Disc Herniation; Lumbar Spinal Stenosis
Keywords: lumbar spine surgery; local anesthesia; local anesthetic block
MeSH Terms: conditions — Spinal Diseases; Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lumbar spine surgery with preoperative fluoroscopically-guided DR block: Patients who have undergone lumbar spine surgery with a fluoroscopically-guided DR block placed by the operative neurosurgeon prior to surgery. These patients subsequently received standard of care general anesthesia and standard multimodality postoperative pain control.
  Interventions: Procedure: Preoperative fluoroscopically-guided dorsal ramus block placed by the operative neurosurgeon
- Lumbar spine surgery without preoperative fluoroscopically-guided DR block: Patients who have undergone lumbar spine surgery without placement of a fluoroscopically-guided DR block. These patients received standard of care general anesthesia and standard multimodality postoperative pain control.

INTERVENTIONS:
Procedure: Preoperative fluoroscopically-guided dorsal ramus block placed by the operative neurosurgeon — Patients received bupivicaine injections delivered via 22-gauge spinal needle to the junction of the facet and transverse process or ala at multiple spinal levels (2.5-5 cc per injection of 0.25% or 0.5% bupivacaine).
  Other Names: Local anesthetic block
  Groups: Lumbar spine surgery with preoperative fluoroscopically-guided DR block

SUMMARY:
The purpose of the this study to evaluate the feasibility, safety, and efficacy of a fluoroscopically-guided dorsal ramus block placed by the operative neurosurgeon prior to lumbosacral surgery. The study will consist of a retrospective analysis of a cohort of patients who underwent lumbosacral surgery patients between June 2018 and March 2021 with or without a preoperative fluoroscopically-guided dorsal ramus (DR) block placed by the operative neurosurgeon.

DETAILED DESCRIPTION:
Spine surgery poses unique challenges in postoperative pain management. Local anesthetic blocks, namely the erector spinae plane and thoracolumbar interfacial plane blocks, placed by anesthesia under ultrasound guidance have been shown to reduce postoperative pain after spinal surgery and decrease perioperative opioid requirements by as much as 50%. Nonetheless these procedures are not routinely performed, likely due to logistical hurdles and lack of widespread knowledge of the procedure by anesthesiologists. A preoperative dorsal ramus block performed by the operative neurosurgeon under fluoroscopy shows promise as an alternative approach to perioperative pain control. The objective of this retrospective observational study is to evaluate the feasibility, safety, and efficacy of a dorsal ramus block block performed by a neurosurgeon under x-ray guidance prior to lumbar surgery. The study will include a cohort of patients who have undergone lumbar spine surgery with or without the x-ray guided dorsal ramus block. A retrospective chart review of these patients will be performed to assess for postoperative pain control, postoperative opioid requirements, time to block completion, length of stay, and adverse events. Descriptive and comparative statistics will be performed. No new data will be gathered from the subjects beyond pre-existing data within the medical record, and no new procedures will be performed as part of the study. If the current study suggests that a dorsal ramus block performed by the operative neurosurgeon is feasible, safe, and effective, it will serve as a foundation for a randomized clinical trial of such a block among patients undergoing lumbar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients undergoing lumbar spine surgery at any spinal level from L1 to sacrum (including decompression, discectomy, posterior fusion, interbody fusion, wound revision or washout, intradural tumor resection, treatment of vascular spinal lesion, tethered cord release, repair of cerebrospinal fluid (CSF) leak, hardware removal)

Exclusion Criteria:

* Patients undergoing surgery that includes thoracic levels
* Patients from whom pain scores could not be elicited in the immediate postoperative period due to mental status (e.g. prolonged intubation requirement, etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population consists of a convenience sample of patients undergoing lumbar spine surgery at a tertiary care academic medical center and an associated specialized spine hospital.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
First visual analog scale (VAS) pain score in the post-anesthesia care unit (PACU) | Within the first 24 hours of surgery
  The first VAS pain score recorded within the PACU on a 0-10 scale, with 0 indicating no pain (better outcome) and 10 indicating more pain (worse outcome).
Total PACU opioid requirements | Within the first 24 hours of surgery
  Total opioids received within the PACU prior to discharge home or transfer to floor (oral morphine equivalents)

SECONDARY OUTCOMES:
Time required to perform block (in minutes) | Up to 30 minutes from start of DR block placement
  Among patients who received DR block, total procedure time required to perform the block, intraoperatively.
Length of Stay (in hours to days) | Up to 30 days from completion of surgery during hospital course
  Total time in hospital from end of surgery to discharge
Total number of adverse events | Up to 24 hours from start of DR block placement
  Adverse cardiovascular events (hypotension, arrhythmia, cardiac arrest), adverse neurological events (unexpected neurological deficit, seizures, changes in intraoperative neuromonitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Christoper E. Mandigo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided